CLINICAL TRIAL: NCT07347899
Title: A Preliminary Study on the Phonetics of Resonance and Articulation Disorders Caused by Defects of the Oral and Maxillofacial Speech Organs and Speech Therapy
Brief Title: Speech-based AI-driven Diagnostics and Rehabilitation for Oral and Oropharyngeal Cancer.
Acronym: speech omics
Status: Completed | Type: Observational
Sponsor: Yudong Xiao (Other)
Responsible Party: Sponsor-Investigator, Yudong Xiao, Dr., Hospital of Stomatology, Sun Yat-Sen University
Organization: Hospital of Stomatology, Sun Yat-Sen University (Other)
Other Study IDs: ERC-[2014]-35
Record Dates: First submitted 2025-12-04; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Oral Cancer; Oropharyngeal Cancer
Keywords: speech signal analysis; diagnostic models; vowel acoustics; bio-inspired computing
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — speech samples will be recorded and saved with anonymization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy control and oral potentially malignant lesion: Speakers with oral potentially malignant lesions or healthy status
- oral cancer and oropharyngeal cancer: Patients diagnosed with oral cancer or oropharyngeal cancer

SUMMARY:
Participants diagnosed with oral cancer, oropharyngeal cancer, or oral potentially malignant lesions, as well as healthy controls, had their speech audio recordings collected for the development and validation of AI-driven models for diagnosis and prognosis prediction of oral cancer and oropharyngeal cancer.

DETAILED DESCRIPTION:
Participants were instructed to articulate three sustained vowels (/a/, /i/, /u/) repeatedly at a moderate volume and pace, with three repetitions per vowel and each utterance lasting at least one second. We developed a neuromorphic computing framework that orthogonally decomposes acoustic features into ultra-dimensional omics representations, enabling the characterization of both localized lesions and systemic physiological conditions. The study collected a comprehensive spectrum of biological profiles, including sociodemographic characteristics, tumor metrics, oral function-related factors, patient-reported outcome measures (PROMs), immunoinflammatory indices, and general health status indicators, to thoroughly investigate the paralinguistic representations of transformed speech omics features. These features were then rigorously evaluated for their clinical efficacy across multiple diagnostic tasks, including screening, early detection, pathological diagnosis, disease staging, and risk factor identification.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as having OC or OPC regardless of concrete pathological subtype (e.g., epithelial, adenoid, odontogenic)
* without a history of other tumor-related treatment before the initial evaluation, such as radiotherapy and chemotherapy
* native Chinese speakers

Exclusion Criteria:

* hearing impairment
* history of stuttering, cerebrovascular accident, brain trauma, neurodegenerative diseases
* severe dental or maxillofacial deformity
* cleft lip, cleft palate, and related post-treatment status
* severe cardiology conditions, breathing/pulmonology disorders, psychiatric disorders or other illnesses preventing patients from receiving standard surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only participants whose self-identified gender aligns with their assigned sex at birth will be included in the study.
Study Population: In-patient participants diagnosed with oral cancer, oropharyngeal cancer or oral potentially malignant lesion and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
AUC value | From enrollment to the report of surgical pathology，up to two weeks.
  Area under the receiver operating characteristic curve (AUC) for discriminating OC/OPC from healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- Department of oral and maxillofacial surgery, Hospital of Stomatology, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Raw audio files and corresponding metadata files for this study are uploaded and shared. The underlying code for this study, including PRAAT scripts for speech preprocessing and automatic feature extraction, and python codes for speech omics representation, can be accessed.
Supporting Information: Analytic Code
Time Frame: permanent valid
URL: https://github.com/Xiaoyud417/SOR